CLINICAL TRIAL: NCT00706446
Title: Genotype Stratified Treatment With Anticholinergic vs. Beta-agonist (Long Acting) and Exacerbations (GABLE)
Brief Title: The Effects of Different Long-acting Bronchodilator Medications on Asthma Patients With Different Genetic Variations
Acronym: GABLE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding was terminated
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Baim Institute for Clinical Research (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Elliot Israel, MD, Director of the Asthma Research Center, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-P-000285
Record Dates: First submitted 2008-06-25; First posted 2008-06-27 (Estimated); Results first posted 2017-05-01 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Asthma
Keywords: Asthma; Pharmacogenetics; Beta agonists; salmeterol; formoterol; tiotropium; beta adrenergic receptor; single nucleotide polymorphism
MeSH Terms: conditions — Asthma | interventions — Tiotropium Bromide; Salmeterol Xinafoate; Formoterol Fumarate; Fluticasone; Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1 - Tio/ICS in the Arg/Arg genotype (Experimental): Tiotropium bromide 18 mcg qd plus inhaled steroids, either Fluticasone propionate Diskus 100 mcg 1 puff bid, Fluticasone propionate aerosol 44 mcg 2 puffs bid, Fluticasone propionate aerosol 110 mcg 2 puffs bid, Fluticasone propionate aerosol 220 mcg 2 puffs qd, Budesonide 90 mcg 2 puffs bid, or Budesonide 180 mcg 2 puffs bid, in the Arg/Arg genotype
  Interventions: Drug: tiotropium bromide; Drug: Fluticasone propionate; Drug: budesonide
- 2 - Tio/ICS in the Arg/Gly genotype (Experimental): Tiotropium bromide 18 mcg QD plus inhaled steroids, either Fluticasone propionate Diskus 100 mcg 1 puff bid, Fluticasone propionate aerosol 44 mcg 2 puffs bid, Fluticasone propionate aerosol 110 mcg 2 puffs bid, Fluticasone propionate aerosol 220 mcg 2 puffs qd, Budesonide 90 mcg 2 puffs bid, or Budesonide 180 mcg 2 puffs bid, in the Arg/Gly genotype
  Interventions: Drug: tiotropium bromide; Drug: Fluticasone propionate; Drug: budesonide
- 3 - Tio/ICS in the Gly/Gly genotype (Experimental): Tiotropium bromide 18 mcg QD plus inhaled steroids, either Fluticasone propionate Diskus 100 mcg 1 puff bid, Fluticasone propionate aerosol 44 mcg 2 puffs bid, Fluticasone propionate aerosol 110 mcg 2 puffs bid, Fluticasone propionate aerosol 220 mcg 2 puffs qd, Budesonide 90 mcg 2 puffs bid, or Budesonide 180 mcg 2 puffs bid, in the Gly/Gly genotype
  Interventions: Drug: tiotropium bromide; Drug: Fluticasone propionate; Drug: budesonide
- 4 - LABA/ICS in the Arg/Arg genotype (Active Comparator): Salmeterol 50 mcg 1 puff BID or Formoterol 12mcg 1 puff BID plus inhaled steroid, either Fluticasone propionate Diskus 100 mcg 1 puff bid, Fluticasone propionate aerosol 44 mcg 2 puffs bid, Fluticasone propionate aerosol 110 mcg 2 puffs bid, Fluticasone propionate aerosol 220 mcg 2 puffs qd, Budesonide 90 mcg 2 puffs bid, or Budesonide 180 mcg 2 puffs bid, in the Arg/Arg genotype
  Interventions: Drug: Salmeterol; Drug: Formoterol; Drug: Fluticasone propionate; Drug: budesonide
- 5 - LABA/ICS in the Arg/Gly genotype (Active Comparator): Salmeterol 50 mcg 1 puff BID or Formoterol 12mcg 1 puff BID plus inhaled steroid, either Fluticasone propionate Diskus 100 mcg 1 puff bid, Fluticasone propionate aerosol 44 mcg 2 puffs bid, Fluticasone propionate aerosol 110 mcg 2 puffs bid, Fluticasone propionate aerosol 220 mcg 2 puffs qd, Budesonide 90 mcg 2 puffs bid, or Budesonide 180 mcg 2 puffs bid, in the Arg/Gly genotype
  Interventions: Drug: Salmeterol; Drug: Formoterol; Drug: Fluticasone propionate; Drug: budesonide
- 6 - LABA/ICS in the Gly/Gly genotype (Active Comparator): Salmeterol 50 mcg 1 puff BID or Formoterol 12mcg 1 puff BID plus inhaled steroid, either Fluticasone propionate Diskus 100 mcg 1 puff bid, Fluticasone propionate aerosol 44 mcg 2 puffs bid, Fluticasone propionate aerosol 110 mcg 2 puffs bid, Fluticasone propionate aerosol 220 mcg 2 puffs qd, Budesonide 90 mcg 2 puffs bid, or Budesonide 180 mcg 2 puffs bid, in the Gly-Gly genotype
  Interventions: Drug: Salmeterol; Drug: Formoterol; Drug: Fluticasone propionate; Drug: budesonide

INTERVENTIONS:
Drug: tiotropium bromide — tiotropium bromide one inhalation a day for one year, along with inhaled steroids at variable dosing based on patient's prior inhaled steroid dosing and treating physician's judgement.
  Other Names: Spiriva
  Arms: 1 - Tio/ICS in the Arg/Arg genotype; 2 - Tio/ICS in the Arg/Gly genotype; 3 - Tio/ICS in the Gly/Gly genotype
Drug: Salmeterol — salmeterol diskus 1 puff twice a day for 1 year, depending on which medication the patient was on before the start of the trial. The goal of this intervention is to continue the patient's current therapy of long-acting beta-agonists. In addition, the patients will be on inhaled steroids at variable doses, depending on what dose they were on at the start of the trial and based on the judgement of their treating physicians.
  Other Names: Serevent
  Arms: 4 - LABA/ICS in the Arg/Arg genotype; 5 - LABA/ICS in the Arg/Gly genotype; 6 - LABA/ICS in the Gly/Gly genotype
Drug: Formoterol — formoterol aerolizer 12 mcg 1 puff twice a day for 1 year, depending on which medication the patient was on before the start of the trial. The goal of this intervention is to continue the patient's current therapy of long-acting beta-agonists. In addition, the patients will be on inhaled steroids at variable doses, depending on what dose they were on at the start of the trial and based on the judgement of their treating physicians.
  Other Names: Foradil
  Arms: 4 - LABA/ICS in the Arg/Arg genotype; 5 - LABA/ICS in the Arg/Gly genotype; 6 - LABA/ICS in the Gly/Gly genotype
Drug: Fluticasone propionate — Either fluticasone propionate diskus 100 mcg 1 puff twice a day or fluticasone propionate aersol in 44 mcg, 110 mcg, 2 puffs twice a day OR fluticasone propionate 220 mcg 2 puffs once a day for one year, depending on which dose the patient was on before the start of the trial.
  Other Names: Flovent
Drug: budesonide — Either budesonide 90 mcg 2 puffs twice a day or 180 mcg 2 puffs twice a day for one year, depending on which dose the patient was on before the start of the trial.
  Other Names: Pulmicort Flexihaler

SUMMARY:
This study is looking at the effects of certain long-acting bronchodilators on patients with asthma who have specific genetic variations. The investigators are interested in a certain common genetic variation in the receptor for beta-agonists, which is found in as many of one-sixth of the population. There is evidence that patients with asthma who have this variation may not do as well when treated with albuterol on a regular basis. The investigators will be looking at whether patients with this variation have more asthma exacerbations over the course of a year when treated with salmeterol or formoterol, which are long-acting forms of albuterol; and whether these patients have fewer exacerbations when treated with tiotropium, which is a different long-acting bronchodilator that does not act at this receptor. In both groups patients will also be receiving inhaled steroids.

DETAILED DESCRIPTION:
Asthma affects 7% of the population in the United States. Asthma morbidity and mortality has increased over the past decade. Long-acting β-agonists (LABAs) combined with inhaled corticosteroids are the most rapidly growing form of asthma therapy in the USA. The only currently USA licensed pharmaceutical that combines a long-acting beta-agonist, salmeterol, and an inhaled corticosteroid is a product know as Advair®. It has become the most widely prescribed asthma controller medication in the United States. While studies have suggested that the combination of a LABA and an inhaled corticosteroid (LABA/ICS), on average, improves asthma control, other studies have suggested that a subpopulation of asthmatics may be at risk for severe exacerbations or death with the use of these agents. These latter studies have caused the FDA to place a "black box" warning on Advair®.

The primary site of therapeutic action of the β-agonists is the beta-adrenergic receptor (ADRB2). One of the common SNPs (allele frequency 0.4 in caucasians) in the coding region of ADRB2 codes for arginine instead of glycine at the 16th amino-acid position of the receptor. In a retrospective association study, we reported that homozygosity for the arginine polymorphism at the 16th amino-acid position (B16 Arg/Arg) as compared to homozygosity for glycine at that position (B16 Gly/Gly) was associated with adverse pulmonary function outcomes when patients used short-acting β-agonists regularly. This report was followed by a study from another group associating increased rates of exacerbations with regular use of short-acting β-agonist in B16 Arg/Arg patients. We subsequently organized and led the first non-oncologic prospective, controlled, double-blinded, genotype stratified trial. In this trial we randomized B16 Arg/Arg and B16 Gly/Gly patients with asthma to regular short-acting β-agonist therapy vs. as needed anti-cholinergic bronchodilator therapy. We showed that patients harboring B16 Arg/Arg, as compared with B16 Gly/Gly, benefited when their use of short-acting β-agonists was minimized by substituting an anti-cholinergic bronchodilator for the β-adrenergic bronchodilator.

Recently, we performed a genotype stratified analysis of patients who had participated in randomized trials using the LABA, salmeterol. We demonstrated that B16 Arg/Arg was associated with adverse outcomes even when the LABA was used with a concomitant inhaled corticosteroid. A recent cross-sectional analysis of pediatric patients using LABAs with ICS suggested that the OR was 3.4 for exacerbations over 6 months in Arg/Arg patients as compared with Gly/Gly patients. In this study, the OR for exacerbation in the presence of the B16 Arg allele in a codominant model was 1.8. Of interest, an industry-sponsored 12 week trial in press did not uncover such an association emphasizing the importance of prospectively confirming these finding[9].

In summary, substantial evidence suggests that asthmatic patients harboring B16 Arg/Arg are at increased risk for adverse outcomes when using a LABA and that they may benefit from the use of an anticholinergic.

A search of the RPDR across all Partners' sites in October 2006, revealed that 13,682 adults age 18-70 with a diagnosis of asthma are receiving a salmeterol containing preparation. At minimum 2.200 of these patients are Arg/Arg (likely more, since the frequency of B16 Arg/Arg is higher in Blacks and Asians). Multiple studies have suggested that patients requiring LABA/ICS therapy experience on average 0.3-0.6 exacerbations per year. The Palmer and Taylor studies suggest that the risk of exacerbations in Arg/Arg patients may be increased from 50-100% by exposure to regular β-agonist therapy. Based on these risks, alternative therapies could potentially reduce the rates of exacerbations by 1/3 to 1/2 in this subpopulation.

We therefore propose a prospective trial in which patients prescribed Advair®, or another combination of a LABA/ICS, are randomized, in a genotype stratified manner, to either continue on therapy with LABA/ICS preparations or to therapy with a long-acting anti-cholinergic/ICS. The primary outcome will be exacerbations as defined by events requiring oral corticosteroids, emergency room visits, or hospitalizations over the one year after randomization[1]. Secondary outcomes will include symptom-free days and quality of life (which we have assessed in prior studies utilizing validated instruments), days lost from work or school, lung function, and non-invasive measures of lung inflammation through collection of exhaled nitric oxide and exhaled breath condensate for assessment of oxidative stress through measures of pH. All techniques and procedures have been utilized by our team at BWH in the course of our prior asthma clinical studies and pharmacogenetic studies.

The primary objective of this study will be address the questions of whether the presence of the arginine polymorphism at the 16th amino-acid of ADRB2 increases the rate of exacerbations in patients with asthma treated with LABA/ICS and whether treatment with an anti-cholinergic/ICS in patients with asthma homozygous for the arginine polymorphism at the 16th amino-acid of ADRB2 reduce exacerbations as compared with treatment with LABA/ICS.

ELIGIBILITY:
Inclusion Criteria:

* Clinical history consistent with asthma
* Has a current prescription for a long-acting beta agonist, either along or in combination with an inhaled corticosteroid (salmeterol, formoterol, fluticasone/salmeterol, or budesonide/formoterol)
* Ability to provide informed consent
* Non-smoker (total lifetime smoking history < 10 pack-years; no more than five occasions of smoking any substance or using smokeless tobacco products in the past year)
* No smoking or use of smokeless tobacco in the past 30 days
* No known contraindication to inhaled tiotropium e.g. narrow angle glaucoma, history of bladder neck obstruction or significant symptoms related to prostatic hypertrophy

Exclusion Criteria:

* Lung disease other than asthma
* Established or suspected diagnosis of vocal cord dysfunction
* Significant medical illness (other than asthma) that is not stable
* History of life-threatening asthma requiring treatment with intubation and mechanical ventilation within the past 5 years
* History of respiratory tract infection within the previous 4 weeks (only applies at screening visits)
* Hyposensitization therapy other than an established maintenance regimen
* Allergy to tiotropium
* Pregnancy or lactation. If potentially able to bear children, not using an acceptable form of birth control
* Inability to use inhaler devices
* Inability to participate over the one year period
* Current use of tiotropium

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2008-06; Primary Completion 2010-06 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Israel, MD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Brigham and Women's Hospital Asthma Research Center — http://www.asthmabwh.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for the GABLE study took place from 06/01/2008 to 06/01/2010 at the Asthma Research Center at Brigham and Women's Hospital.
Groups:
- 1 - Tiotropium Plus ICS in the Arg/Arg Genotype: Tiotropium bromide 18 mcg qd plus inhaled steroids, either Fluticasone propionate Diskus 100 mcg 1 puff bid, Fluticasone propionate aerosol 44 mcg 2 puffs bid, Fluticasone propionate aerosol 110 mcg 2 puffs bid, Fluticasone propionate aerosol 220 mcg 2 puffs qd, Budesonide 90 mcg 2 puffs bid, or Budesonide 180 mcg 2 puffs bid, in the Arg/Arg genotype
  tiotropium bromide: tiotropium bromide one inhalation a day for one year
  Fluticasone propionate: Either fluticasone propionate diskus 100 mcg 1 puff twice a day or fluticasone propionate aersol in 44 mcg, 110 mcg, 2 puffs twice a day OR fluticasone propionate 220 mcg 2 puffs once a day for one year, dosing based on patient's prior inhaled steroid dosing and treating physician's judgement.
  budesonide: Either budesonide 90 mcg 2 puffs twice a day or 180 mcg 2 puffs twice a day for one year, ddosing based on patient's prior inhaled steroid dosing and treating physician's judgement.
- 2 - Tiotropium Plus ICS in the Arg/Gly Genotype: Tiotropium bromide 18 mcg QD plus inhaled steroids, either Fluticasone propionate Diskus 100 mcg 1 puff bid, Fluticasone propionate aerosol 44 mcg 2 puffs bid, Fluticasone propionate aerosol 110 mcg 2 puffs bid, Fluticasone propionate aerosol 220 mcg 2 puffs qd, Budesonide 90 mcg 2 puffs bid, or Budesonide 180 mcg 2 puffs bid, in the Arg/Gly genotype
  tiotropium bromide: tiotropium bromide one inhalation a day for one year
  Fluticasone propionate: Either fluticasone propionate diskus 100 mcg 1 puff twice a day or fluticasone propionate aersol in 44 mcg, 110 mcg, 2 puffs twice a day OR fluticasone propionate 220 mcg 2 puffs once a day for one year, dosing based on patient's prior inhaled steroid dosing and treating physician's judgement.
  budesonide: Either budesonide 90 mcg 2 puffs twice a day or 180 mcg 2 puffs twice a day for one year, dosing based on patient's prior inhaled steroid dosing and treating physician's judgement.
- 3 - Tiotropium Plus ICS in the Gly/Gly Genotype: Tiotropium bromide 18 mcg QD plus inhaled steroids, either Fluticasone propionate Diskus 100 mcg 1 puff bid, Fluticasone propionate aerosol 44 mcg 2 puffs bid, Fluticasone propionate aerosol 110 mcg 2 puffs bid, Fluticasone propionate aerosol 220 mcg 2 puffs qd, Budesonide 90 mcg 2 puffs bid, or Budesonide 180 mcg 2 puffs bid, in the Gly/Gly genotype
  tiotropium bromide: tiotropium bromide one inhalation a day for one year
  Fluticasone propionate: Either fluticasone propionate diskus 100 mcg 1 puff twice a day or fluticasone propionate aersol in 44 mcg, 110 mcg, 2 puffs twice a day OR fluticasone propionate 220 mcg 2 puffs once a day for one year, dosing based on patient's prior inhaled steroid dosing and treating physician's judgement.
  budesonide: Either budesonide 90 mcg 2 puffs twice a day or 180 mcg 2 puffs twice a day for one year, dosing based on patient's prior inhaled steroid dosing and treating physician's judgement.p
- 4 - Salmeterol or Formoterol Plus ICS in the Arg/Arg Genotype: Salmeterol 50 mcg 1 puff BID or Formoterol 12mcg 1 puff BID plus inhaled steroid, either Fluticasone propionate Diskus 100 mcg 1 puff bid, Fluticasone propionate aerosol 44 mcg 2 puffs bid, Fluticasone propionate aerosol 110 mcg 2 puffs bid, Fluticasone propionate aerosol 220 mcg 2 puffs qd, Budesonide 90 mcg 2 puffs bid, or Budesonide 180 mcg 2 puffs bid, in the Arg/Arg genotype
  Salmeterol: salmeterol diskus 1 puff twice a day for 1 year OR
  Formoterol: formoterol aerolizer 12 mcg 1 puff twice a day for 1 year, depending on which medication the patient was on before the start of the trial.
  Fluticasone propionate: Either fluticasone propionate diskus 100 mcg 1 puff twice a day or fluticasone propionate aersol in 44 mcg, 110 mcg, 2 puffs twice a day OR fluticasone propionate 220 mcg 2 puffs once a day for one year,
  OR budesonide: Either budesonide 90 mcg 2 puffs twice a day or 180 mcg 2 puffs twice a day for one year. Dosing based on patient's prior inhaled steroid dosing.
- 5 - Salmeterol or Formoterol Plus ICS in the Arg/Gly Genotype: Salmeterol 50 mcg 1 puff BID or Formoterol 12mcg 1 puff BID plus inhaled steroid, either Fluticasone propionate Diskus 100 mcg 1 puff bid, Fluticasone propionate aerosol 44 mcg 2 puffs bid, Fluticasone propionate aerosol 110 mcg 2 puffs bid, Fluticasone propionate aerosol 220 mcg 2 puffs qd, Budesonide 90 mcg 2 puffs bid, or Budesonide 180 mcg 2 puffs bid, in the Arg-Gly genotype
  Salmeterol: salmeterol diskus 1 puff twice a day for 1 year OR
  Formoterol: formoterol aerolizer 12 mcg 1 puff twice a day for 1 year, depending on which medication the patient was on before the start of the trial.
  Fluticasone propionate: Either fluticasone propionate diskus 100 mcg 1 puff twice a day or fluticasone propionate aersol in 44 mcg, 110 mcg, 2 puffs twice a day OR fluticasone propionate 220 mcg 2 puffs once a day for one year,
  OR budesonide: Either budesonide 90 mcg 2 puffs twice a day or 180 mcg 2 puffs twice a day for one year. Dosing based on patient's prior inhaled steroid dosing.
- 6 - Salmeterol or Formoterol Plus ICS in the Gly/Gly Genotype: Salmeterol 50 mcg 1 puff BID or Formoterol 12mcg 1 puff BID plus inhaled steroid, either Fluticasone propionate Diskus 100 mcg 1 puff bid, Fluticasone propionate aerosol 44 mcg 2 puffs bid, Fluticasone propionate aerosol 110 mcg 2 puffs bid, Fluticasone propionate aerosol 220 mcg 2 puffs qd, Budesonide 90 mcg 2 puffs bid, or Budesonide 180 mcg 2 puffs bid, in the Gly-Gly genotype
  Salmeterol: salmeterol diskus 1 puff twice a day for 1 year OR
  Formoterol: formoterol aerolizer 12 mcg 1 puff twice a day for 1 year, depending on which medication the patient was on before the start of the trial.
  Fluticasone propionate: Either fluticasone propionate diskus 100 mcg 1 puff twice a day or fluticasone propionate aersol in 44 mcg, 110 mcg, 2 puffs twice a day OR fluticasone propionate 220 mcg 2 puffs once a day for one year,
  OR budesonide: Either budesonide 90 mcg 2 puffs twice a day or 180 mcg 2 puffs twice a day for one year. Dosing based on patient's prior inhaled steroid dosing.
Period: Overall Study
Arm/Group | 1 - Tiotropium Plus ICS in the Arg/Arg Genotype | 2 - Tiotropium Plus ICS in the Arg/Gly Genotype | 3 - Tiotropium Plus ICS in the Gly/Gly Genotype | 4 - Salmeterol or Formoterol Plus ICS in the Arg/Arg Genotype | 5 - Salmeterol or Formoterol Plus ICS in the Arg/Gly Genotype | 6 - Salmeterol or Formoterol Plus ICS in the Gly/Gly Genotype
Started | 29 | 57 | 44 | 26 | 54 | 45
Completed | 3 | 8 | 7 | 4 | 10 | 7
Not Completed | 26 | 49 | 37 | 22 | 44 | 38

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 - Tiotropium Plus ICS in the Arg/Arg Genotype | 2 - Tiotropium Plus ICS in the Arg/Gly Genotype | 3 - Tiotropium Plus ICS in the Gly/Gly Genotype | 4 - Salmeterol or Formoterol Plus ICS in the Arg/Arg Genotype | 5 - Salmeterol or Formoterol Plus ICS in the Arg/Gly Genotype | 6 - Salmeterol or Formoterol Plus ICS in the Gly/Gly Genotype | Total
Number analyzed (Participants) | 29 | 57 | 44 | 26 | 54 | 45 | 255
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One participant is missing information on age in the Salmeterol or Formoterol plus ICS in the Arg/Arg genotype group.
  years
    number analyzed (Participants) | 29 | 57 | 44 | 25 | 54 | 45 | 254
    (all) | 47.3 (15.9) | 45.7 (13.2) | 46.0 (16.3) | 46.6 (14.2) | 50.3 (14.7) | 50.5 (13.6) | 47.85 (14.58)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One participant in the Salmeterol or Formoterol plus ICS in the Arg/Gly genotype group is missing sex information.
  Participants
    number analyzed (Participants) | 29 | 57 | 44 | 26 | 53 | 45 | 254
    Female | 8 | 14 | 14 | 8 | 21 | 11 | 76
    Male | 21 | 43 | 30 | 18 | 32 | 34 | 178
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 57 | 44 | 26 | 54 | 45 | 255

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Asthma Exacerbation
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | 1 - Tiotropium Plus ICS in the Arg/Arg Genotype | 2 - Tiotropium Plus ICS in the Arg/Gly Genotype | 3 - Tiotropium Plus ICS in the Gly/Gly Genotype | 4 - Salmeterol or Formoterol Plus ICS in the Arg/Arg Genotype | 5 - Salmeterol or Formoterol Plus ICS in the Arg/Gly Genotype | 6 - Salmeterol or Formoterol Plus ICS in the Gly/Gly Genotype
Number analyzed (Participants) | 29 | 57 | 44 | 26 | 54 | 45
Participants | 3 | 15 | 6 | 6 | 12 | 9

2. Secondary Outcome: FEV1 (Forced Expiratory Volume)
Time Frame: 1 year
Population: Data was not collected for secondary outcomes due to study termination
Arm/Group | 1 - Tiotropium Plus ICS in the Arg/Arg Genotype | 2 - Tiotropium Plus ICS in the Arg/Gly Genotype | 3 - Tiotropium Plus ICS in the Gly/Gly Genotype | 4 - Salmeterol or Formoterol Plus ICS in the Arg/Arg Genotype | 5 - Salmeterol or Formoterol Plus ICS in the Arg/Gly Genotype | 6 - Salmeterol or Formoterol Plus ICS in the Gly/Gly Genotype
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Exhaled NO (Nitric Oxide)
Time Frame: 1 year
Population: Data was not collected for secondary outcomes due to study termination.
Arm/Group | 1 - Tiotropium Plus ICS in the Arg/Arg Genotype | 2 - Tiotropium Plus ICS in the Arg/Gly Genotype | 3 - Tiotropium Plus ICS in the Gly/Gly Genotype | 4 - Salmeterol or Formoterol Plus ICS in the Arg/Arg Genotype | 5 - Salmeterol or Formoterol Plus ICS in the Arg/Gly Genotype | 6 - Salmeterol or Formoterol Plus ICS in the Gly/Gly Genotype
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Symptom-free Days
Time Frame: 1 year
Population: Data was not collected for secondary outcomes due to study termination.
Arm/Group | 1 - Tiotropium Plus ICS in the Arg/Arg Genotype | 2 - Tiotropium Plus ICS in the Arg/Gly Genotype | 3 - Tiotropium Plus ICS in the Gly/Gly Genotype | 4 - Salmeterol or Formoterol Plus ICS in the Arg/Arg Genotype | 5 - Salmeterol or Formoterol Plus ICS in the Arg/Gly Genotype | 6 - Salmeterol or Formoterol Plus ICS in the Gly/Gly Genotype
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Asthma-related Quality of Life
Time Frame: 1 year
Population: Data was not collected for secondary outcomes due to study termination.
Arm/Group | 1 - Tiotropium Plus ICS in the Arg/Arg Genotype | 2 - Tiotropium Plus ICS in the Arg/Gly Genotype | 3 - Tiotropium Plus ICS in the Gly/Gly Genotype | 4 - Salmeterol or Formoterol Plus ICS in the Arg/Arg Genotype | 5 - Salmeterol or Formoterol Plus ICS in the Arg/Gly Genotype | 6 - Salmeterol or Formoterol Plus ICS in the Gly/Gly Genotype
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: This trial did not collect adverse event data.
Groups:
- 1 - Tio/ICS in the Arg/Arg Genotype: Tiotropium bromide 18 mcg qd plus inhaled steroids, either Fluticasone propionate Diskus 100 mcg 1 puff bid, Fluticasone propionate aerosol 44 mcg 2 puffs bid, Fluticasone propionate aerosol 110 mcg 2 puffs bid, Fluticasone propionate aerosol 220 mcg 2 puffs qd, Budesonide 90 mcg 2 puffs bid, or Budesonide 180 mcg 2 puffs bid, in the Arg/Arg genotype
  tiotropium bromide: tiotropium bromide one inhalation a day for one year, along with inhaled steroids at variable dosing based on patient's prior inhaled steroid dosing and treating physician's judgement.
  Fluticasone propionate: Either fluticasone propionate diskus 100 mcg 1 puff twice a day or fluticasone propionate aersol in 44 mcg, 110 mcg, 2 puffs twice a day OR fluticasone propionate 220 mcg 2 puffs once a day for one year, depending on which dose the patient was on before the start of the trial.
  budesonide: Either budesonide 90 mcg 2 puffs twice a day or 180 mcg 2 puffs twice a day for one year, depending on which dose the p
- 2 - Tio/ICS in the Arg/Gly Genotype: Tiotropium bromide 18 mcg QD plus inhaled steroids, either Fluticasone propionate Diskus 100 mcg 1 puff bid, Fluticasone propionate aerosol 44 mcg 2 puffs bid, Fluticasone propionate aerosol 110 mcg 2 puffs bid, Fluticasone propionate aerosol 220 mcg 2 puffs qd, Budesonide 90 mcg 2 puffs bid, or Budesonide 180 mcg 2 puffs bid, in the Arg/Gly genotype tiotropium bromide: tiotropium bromide one inhalation a day for one year, along with inhaled steroids at variable dosing based on patient's prior inhaled steroid dosing and treating physician's judgement.
  Fluticasone propionate: Either fluticasone propionate diskus 100 mcg 1 puff twice a day or fluticasone propionate aersol in 44 mcg, 110 mcg, 2 puffs twice a day OR fluticasone propionate 220 mcg 2 puffs once a day for one year, depending on which dose the patient was on before the start of the trial.
  budesonide: Either budesonide 90 mcg 2 puffs twice a day or 180 mcg 2 puffs twice a day for one year, depending on which dose the p
- 3 - Tio/ICS in the Gly/Gly Genotype: Tiotropium bromide 18 mcg QD plus inhaled steroids, either Fluticasone propionate Diskus 100 mcg 1 puff bid, Fluticasone propionate aerosol 44 mcg 2 puffs bid, Fluticasone propionate aerosol 110 mcg 2 puffs bid, Fluticasone propionate aerosol 220 mcg 2 puffs qd, Budesonide 90 mcg 2 puffs bid, or Budesonide 180 mcg 2 puffs bid, in the Gly/Gly genotype tiotropium bromide: tiotropium bromide one inhalation a day for one year, along with inhaled steroids at variable dosing based on patient's prior inhaled steroid dosing and treating physician's judgement.
  Fluticasone propionate: Either fluticasone propionate diskus 100 mcg 1 puff twice a day or fluticasone propionate aersol in 44 mcg, 110 mcg, 2 puffs twice a day OR fluticasone propionate 220 mcg 2 puffs once a day for one year, depending on which dose the patient was on before the start of the trial.
  budesonide: Either budesonide 90 mcg 2 puffs twice a day or 180 mcg 2 puffs twice a day for one year, depending on which dose the p
- 4 - LABA/ICS in the Arg/Arg Genotype: Salmeterol 50 mcg 1 puff BID or Formoterol 12mcg 1 puff BID plus inhaled steroid, either Fluticasone propionate Diskus 100 mcg 1 puff bid, Fluticasone propionate aerosol 44 mcg 2 puffs bid, Fluticasone propionate aerosol 110 mcg 2 puffs bid, Fluticasone propionate aerosol 220 mcg 2 puffs qd, Budesonide 90 mcg 2 puffs bid, or Budesonide 180 mcg 2 puffs bid, in the Arg/Arg genotype Salmeterol: salmeterol diskus 1 puff twice a day for 1 year, depending on which medication the patient was on before the start of the trial. The goal of this intervention is to continue the patient's current therapy of long-acting beta-agonists. In addition, the patients will be on inhaled steroids at variable doses, depending on what dose they were on at the start of the trial and based on the judgement of their treating physicians.
  Formoterol: formoterol aerolizer 12 mcg 1 puff twice a day for 1 year, depending on which medication the patient was on before the start of the trial. The goal of this in
- 5 - LABA/ICS in the Arg/Gly Genotype: Salmeterol 50 mcg 1 puff BID or Formoterol 12mcg 1 puff BID plus inhaled steroid, either Fluticasone propionate Diskus 100 mcg 1 puff bid, Fluticasone propionate aerosol 44 mcg 2 puffs bid, Fluticasone propionate aerosol 110 mcg 2 puffs bid, Fluticasone propionate aerosol 220 mcg 2 puffs qd, Budesonide 90 mcg 2 puffs bid, or Budesonide 180 mcg 2 puffs bid, in the Arg/Gly genotype Salmeterol: salmeterol diskus 1 puff twice a day for 1 year, depending on which medication the patient was on before the start of the trial. The goal of this intervention is to continue the patient's current therapy of long-acting beta-agonists. In addition, the patients will be on inhaled steroids at variable doses, depending on what dose they were on at the start of the trial and based on the judgement of their treating physicians.
  Formoterol: formoterol aerolizer 12 mcg 1 puff twice a day for 1 year, depending on which medication the patient was on before the start of the trial. The goal of this in
- 6 - LABA/ICS in the Gly/Gly Genotype: Salmeterol 50 mcg 1 puff BID or Formoterol 12mcg 1 puff BID plus inhaled steroid, either Fluticasone propionate Diskus 100 mcg 1 puff bid, Fluticasone propionate aerosol 44 mcg 2 puffs bid, Fluticasone propionate aerosol 110 mcg 2 puffs bid, Fluticasone propionate aerosol 220 mcg 2 puffs qd, Budesonide 90 mcg 2 puffs bid, or Budesonide 180 mcg 2 puffs bid, in the Gly-Gly genotype Salmeterol: salmeterol diskus 1 puff twice a day for 1 year, depending on which medication the patient was on before the start of the trial. The goal of this intervention is to continue the patient's current therapy of long-acting beta-agonists. In addition, the patients will be on inhaled steroids at variable doses, depending on what dose they were on at the start of the trial and based on the judgement of their treating physicians.
  Formoterol: formoterol aerolizer 12 mcg 1 puff twice a day for 1 year, depending on which medication the patient was on before the start of the trial. The goal of this in
Arm/Group | 1 - Tio/ICS in the Arg/Arg Genotype | 2 - Tio/ICS in the Arg/Gly Genotype | 3 - Tio/ICS in the Gly/Gly Genotype | 4 - LABA/ICS in the Arg/Arg Genotype | 5 - LABA/ICS in the Arg/Gly Genotype | 6 - LABA/ICS in the Gly/Gly Genotype
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No